CLINICAL TRIAL: NCT04052516
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of NST-4016 in Patients With Nonalcoholic Steatohepatitis (NASH)
Brief Title: A Phase 2b Study of Icosabutate in Fatty Liver Disease
Acronym: ICONA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NorthSea Therapeutics B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NST-02
Record Dates: First submitted 2019-08-07; First posted 2019-08-09 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Non Alcoholic Steatohepatitis (NASH)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — icosabutate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo oral capsules taken one daily for 52 weeks
  Interventions: Drug: Placebo
- Icosabutate 300mg (Experimental): Icosabutate 300mg oral capsule taken once daily for 52 weeks
  Interventions: Drug: Icosabutate
- Icosabutate 600mg (Experimental): Icosabutate 600mg oral capsules taken once daily for 52 weeks
  Interventions: Drug: Icosabutate

INTERVENTIONS:
Drug: Icosabutate — Icosabutate oral capsule once daily
  Other Names: NST-4016
  Arms: Icosabutate 300mg; Icosabutate 600mg
Drug: Placebo — Matching placebo oral capsule
  Arms: Placebo

SUMMARY:
A Phase 2b study to evaluate the efficacy of different doses of NST-4016 on the resolution of NASH without worsening of fibrosis

DETAILED DESCRIPTION:
This is a 62 week (including screening and follow-up), multicenter, randomized, double blind, placebo-controlled, parallel group study in male and female patients with a histological diagnosis of NASH. The study includes a screening period, double blind treatment period, and post-treatment follow up

ELIGIBILITY:
Inclusion Criteria:

* Provides signed written informed consent and agrees to comply with the study protocol.
* Is a male or female aged 18 to 75 years, inclusive.
* Has a histological diagnosis of NASH prior to study entry
* Has (NAS) greater than or equal to 4, with a score of at least 1 in each component (steatosis, lobular inflammation, and ballooning),
* Has a fibrosis score F1 to F3, inclusive (F1 capped at 30%),
* Has a Proton Density Fat Fraction (PDFF) greater than or equal to 10% on MRI at screening

Exclusion Criteria:

* Has a known history of alcohol abuse or daily heavy alcohol consumption
* Has had bariatric surgery within the past 5 years
* Has significant systemic or major illnesses other than liver disease
* Has a recent (within 6 months) history of cardiac dysrhythmias and/or cardiovascular disease
* Has uncontrolled arterial hypertension
* Positive for Hep B, Hepatitis C Virus (HCV) or HCV Polymerase Chain Reaction (PCR)
* Has type 1 diabetes mellitus
* Has diabetic ketoacidosis
* Has a history of liver decompensation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2019-07-17 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-12-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (38):
  - Central ResearchAssociates Inc., Birmingham, Alabama
  - Arizona Liver Health, Chandler, Arizona
  - Arizona Liver Health - Glendale, Glendale, Arizona
  - Arizona Liver Health, Tucson, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Arkansas Gastroenterology - North Little Rock, North Little Rock, Arkansas
  - Fresno Clinical Research Center, Fresno, California
  - National Research Institute - Huntington Park, Huntington Park, California
  - National Research Institute - Wilshire, Los Angeles, California
  - National Research Institute - Panorama, Panorama City, California
  - Alliance Clinical Research, Poway, California
  - National Research Institute - Santa Ana, Santa Ana, California
  - South Denver Gastroenterology, Englewood, Colorado
  - Excel Medical Clinical Trials, LLC, Boca Raton, Florida
  - Sensible Healthcare LLC, Ocoee, Florida
  - Covenant Research LLC, Sarasota, Florida
  - Gastrointestinal Specialists of Georgia PC, Marietta, Georgia
  - University of Chicago, Chicago, Illinois
  - Texas Digestive Disease Consultants, Baton Rouge, Louisiana
  - Tandem Clinical Research, Marrero, Louisiana
  - Gastrointestinal Associates, PA, Flowood, Mississippi
  - Southern Therapy and Advanced Research LLC, Jackson, Mississippi
  - Kansas City Research Institute, Kansas City, Missouri
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - Aventiv Research, Inc., Columbus, Ohio
  - Premier Research, Clarksville, Tennessee
  - Gastro One, Germantown, Tennessee
  - Pinnacle Clinical Research, Austin, Texas
  - Texas Digestive Disease Consultants, Dallas, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Liver Associates of Texas, Houston, Texas
  - Doctors Hospital at Renaissance, LLC, McAllen, Texas
  - Quality Research Inc, San Antonio, Texas
  - American Research Corporation, San Antonio, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Brooke Army Medical Center, San Antonio, Texas
  - Texas Digestive Disease Consultants - Webster, Webster, Texas
  - Hunter Holmes McGuire VA Medical Center, Richmond, Virginia
- Fundacion de Investigacion (FDI), San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrison SA, Alkhouri N, Ortiz-Lasanta G, Rudraraju M, Tai D, Wack K, Shah A, Besuyen R, Steineger HH, Fraser DA, Sanyal AJ; ICONA Study Investigators. A phase IIb randomised-controlled trial of the FFAR1/FFAR4 agonist icosabutate in MASH. J Hepatol. 2025 Aug;83(2):293-303. doi: 10.1016/j.jhep.2025.01.032. Epub 2025 Feb 10. PMID 39938653

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Started | 92 | 93 | 95
Safety Population | 91 | 92 | 95
ITT (The Intent-to-Treat Population included all patients who were randomized and received at least 1 dose of study drug.) | 91 | 92 | 95
mITT (Modified Intent-To-Treat Population - The mITT population included all patients from the ITT Population who had valid baseline and Week 52 (or ET, if applicable) liver biopsy measurements; a valid Week 52/ET liver biopsy was defined as a liver biopsy that had occurred within 90 days of last dose/Week 52 visit.) | 75 | 76 | 77
3-Panel mITT (The 3-Panel mITT Population included all patients who had a baseline and Week 52 (or ET, if applicable) liver biopsy read and fulfilled eligibility criteria based on the 3-panel read paradigm. This population was considered the primary population for the efficacy analysis of the histology data.) | 75 | 76 | 77
Completed | 79 | 78 | 78
Not Completed | 13 | 15 | 17
Not completed — Withdrawal by Subject | 4 | 5 | 6
Not completed — Adverse Event | 3 | 2 | 8
Not completed — Lost to Follow-up | 2 | 5 | 3
Not completed — Protocol Violation | 1 | 1 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Pregnancy | 1 | 0 | 0
Not completed — Requirement of prohibited concomitant medication | 1 | 0 | 0
Not completed — Reason not recorded | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Modified Intent-To-Treat (mITT) Population is used for the baseline analysis population as this was the primary population for efficacy analysis. The mITT Population included all patients from the ITT Population who had valid baseline and Week 52 (or ET, if applicable) liver biopsy measurements; a valid Week 52/ET liver biopsy was defined as a liver biopsy that had occurred within 90 days of last dose/Week 52 visit.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg | Total
Number analyzed (Participants) | 75 | 76 | 77 | 228
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (11.15) | 53.3 (10.52) | 51.8 (10.26) | 53.0 (10.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52 | 55 | 51 | 158
  Male | 23 | 21 | 26 | 70
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 31 | 29 | 92
  Not Hispanic or Latino | 42 | 44 | 45 | 131
  Unknown or Not Reported | 1 | 1 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 1 | 3
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 2 | 5 | 8
  White | 72 | 72 | 71 | 215
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 0 | 1
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 35.94 (6.230) | 36.73 (5.732) | 37.32 (6.047) | 36.67 (6.006)
Alcohol use [Count of Participants; unit: Participants]
  Current | 44 | 40 | 40 | 124
  Former | 10 | 8 | 12 | 30
  Never | 20 | 28 | 25 | 73
  Missing | 1 | 0 | 0 | 1
Type 2 Diabetes status [Count of Participants; unit: Participants]
  Diabetic | 35 | 40 | 39 | 114
  Non-diabetic | 40 | 36 | 38 | 114

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Resolution of NASH, Defined as Disappearance of Ballooning (Score = 0) With Lobular Inflammation Score 0 or 1, With no Worsening of Fibrosis.
Time Frame: 52 weeks
Population: 3-Panel Modified Intent-To-Treat (mITT) Population - The 3-Panel mITT Population included all patients who had a baseline and Week 52 (or ET, if applicable) liver biopsy read and fulfilled eligibility criteria based on the 3-panel read paradigm. This population was considered the primary population for the efficacy analysis of the histology data.
  Biopsy fibrosis score F2/F3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 46 | 52 | 53
percentage of participants | 8.7 | 17.3 | 20.8
Statistical Analysis 1: Comparison: Placebo vs Icosabutate 300mg; Test type: Other — Cochran-Mantel-Haenszal test; p = 0.2991, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.70, 95% CI 2-sided [0.62 to 4.63]
Statistical Analysis 2: Comparison: Placebo vs Icosabutate 600mg; Test type: Other — Cochran-Mantel-Haenszel Test; p = 0.1386, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.01, 95% CI 2-sided [0.80 to 5.08]

2. Secondary Outcome: Percentage of Patients With Fibrosis Improvement, Defined as Greater Than or Equal to 1 Stage of Fibrosis Improvement and no Worsening of Steatohepatitis (Inflammation/Ballooning).
Time Frame: 52 weeks
Population: 3-Panel mITT population. Biopsy fibrosis score F2/F3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 46 | 52 | 53
percentage of participants | 13.0 | 26.9 | 24.5

3. Secondary Outcome: Percentage of Patients With Fibrosis Improvement, Defined as Greater Than or Equal to 1 Stage of Fibrosis Improvement.
Time Frame: 52 weeks
Population: 3-Panel mITT population. Biopsy fibrosis score F2/F3.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 46 | 52 | 53
percentage of participants | 13.0 | 30.8 | 28.3

4. Secondary Outcome: Changes in the Liver Enzymes Aspartate Aminotransferase (AST)U/L, Alanine Aminotransferase ( ALT)U/L and Gamma Glutamyl Transferase (GGT) U/L From Baseline
Time Frame: 52 weeks
Population: Results are presented for those participants in the 3-panel mITT population who had results for these parameters at Week 52.
Measure: Least Squares Mean (Standard Error); unit: U/L
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 61 | 56 | 66
U/L
  Aspartate Aminotransferase | -8.2 (3.18) | -14.9 (3.46) | -18.5 (3.13)
  Alanine Aminotransferase | -9.8 (3.73) | -27.9 (4.05) | -30.1 (3.65)
  Gamma Glutamyl Transferase | -5.1 (5.41) | -27.9 (5.75) | -32.7 (5.26)

5. Secondary Outcome: Change in Bilirubin Micromol/L From Baseline
Time Frame: 52 weeks
Population: Results are presented for those participants in the 3-panel mITT population who had results for this parameter at Week 52
Measure: Least Squares Mean (Standard Error); unit: micromol/L
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 61 | 56 | 66
micromol/L | 0.56 (0.332) | -1.11 (0.362) | -1.49 (0.325)

6. Secondary Outcome: Change From Baseline in Inflammation Marker hsCRP
Time Frame: 52 weeks
Population: 3-panel mITT population
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 62 | 58 | 67
mg/L | 1.089 (0.8095) | -1.297 (0.8953) | -3.382 (0.7978)

7. Secondary Outcome: Change From Baseline in Fibrosis Activity Marker Pro-C3
Time Frame: 52 weeks
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: micrograms/L
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 60 | 54 | 64
micrograms/L | -4.33 (2.830) | -3.68 (3.023) | -11.76 (2.762)

8. Secondary Outcome: Change From Baseline in Fibrosis Activity Marker Enhanced Liver Fibrosis (ELF) Test
Description: ELF is a blood test that measures liver fibrosis by analyzing three markers in the blood: Hyaluronic acid (HA), Procollagen III amino-terminal peptide (PIIINP), and Tissue inhibitor of matrix metalloproteinase 1 (TIMP-1). The higher the score the higher the levels of markers in the blood. ELF score = 2.278 + 0.851 × ln(HA) + 0.751 × ln(PIIINP) + 0.394 × ln(TIMP-1). As the score is a composite measure of the levels of three markers in the blood, there is not a finite range for this parameter.
Time Frame: 52 weeks
Population: as for outcome 4
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 60 | 54 | 64
score | -0.051 (0.0993) | -0.125 (0.1087) | -0.370 (0.0983)

9. Secondary Outcome: Change From Baseline in Homeostasis Model Assessment of Insulin Resistance (HOMA-IR)
Description: HOMA-IR is a measure of insulin resistance and metabolic status. The higher the score, the higher the level of insulin resistance. HOMA-IR = fasting glucose [mmol/L)] × fasting insulin [mIU/L]/22.5. As HOMA-IR is a composite score using 2 parameters, it does not have a finite range.
Time Frame: 52 weeks
Population: 3-panel mITT population
Measure: Least Squares Mean (Standard Error); unit: score
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 62 | 58 | 67
score | 0.609 (1.3453) | -2.810 (1.4733) | -3.794 (1.3203)

10. Secondary Outcome: Change From Baseline in Composite Disease Activity Score (Composite NASH Score of Inflammation, Ballooning, Fibrosis)
Description: The disease activity score can range from 0 to 8 and is calculated by the sum of scores of steatosis (0-3), lobular inflammation (0-3) and hepatocyte ballooning (0-2). The higher the score the more severe the disease.
Time Frame: 52 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 61 | 58 | 66
score on a scale | -0.2 (1.68) | -0.7 (1.84) | -0.9 (1.56)

11. Secondary Outcome: Change From Baseline in Nonalcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS)
Description: A histological scoring system that assesses a liver biopsy and gives scores for steatosis (0-3), lobular inflammation (0-3), and hepatocyte ballooning (0-2) giving a total score of (0-8). The higher the score the more severe the disease
Time Frame: 52 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 61 | 58 | 65
score on a scale | -0.9 (1.36) | -0.9 (1.51) | -1.3 (1.65)

12. Secondary Outcome: Changes in Individual Histological Scores for Steatosis, Ballooning, Inflammation, and Fibrosis From Baseline
Description: Changes in scores for the individual component parts of the Nonalcoholic fatty liver disease (NAFLD) activity score (NAS) as judged by a pathologist examining sections from a liver biopsy; steatosis (range 0-3), lobular inflammation (range 0-3), and hepatocyte ballooning (range 0-2) In all cases a higher number denotes more severe disease activity
Time Frame: 52 weeks
Population: 3-panel mITT population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 62 | 58 | 67
score on a scale
  Steatosis grade: number analyzed (Participants) | 61 | 58 | 65
  Steatosis grade | -0.4 (0.62) | -0.2 (0.65) | -0.4 (0.81)
  Lobular inflammation score: number analyzed (Participants) | 61 | 58 | 67
  Lobular inflammation score | -0.2 (0.62) | -0.4 (0.67) | -0.5 (0.61)
  Hepatocyte ballooning score | -0.3 (0.79) | -0.3 (0.84) | -0.4 (0.78)

13. Secondary Outcome: Change From Baseline in Magnetic Resonance Imaging-Proton Density-Fat Fraction (MRI-PDFF)
Description: MRI-PDFF is a quantitative imaging biomarker that measures the fat fraction of tissue by correcting factors influencing magnetic resonance signal intensity.
Time Frame: 52 weeks
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of fat
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
Number analyzed (Participants) | 62 | 58 | 65
Percentage of fat | -4.37 (7.185) | -1.33 (5.356) | -0.95 (8.206)

ADVERSE EVENTS:
Time Frame: AEs, which included clinical laboratory test variables, were monitored and documented from the time the patient signed the ICF until Visit 10 (Week 54) or the Early Termination visit (if applicable).
Arm/Group | Placebo | Icosabutate 300mg | Icosabutate 600mg
All-Cause Mortality (participants affected / at risk) | 1/91 | 0/92 | 1/95
Serious Adverse Events (participants affected / at risk) | 4/91 | 5/92 | 8/95
Other Adverse Events (participants affected / at risk) | 82/91 | 80/92 | 80/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | Icosabutate 300mg (N=92) | Icosabutate 600mg (N=95)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Coronavirus infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal hematoma (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Transient ischemic attack (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Food allergy (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Post-procedural hematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Coronavirus test positive (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=91) | Icosabutate 300mg (N=92) | Icosabutate 600mg (N=95)
Diarrhea (Gastrointestinal disorders) | 13 (13) | 13 (14) | 15 (17)
Nausea (Gastrointestinal disorders) | 4 (6) | 13 (14) | 22 (24)
Abdominal pain upper (Gastrointestinal disorders) | 3 (4) | 5 (5) | 9 (10)
Abdominal pain (Gastrointestinal disorders) | 6 (6) | 5 (5) | 3 (3)
Constipation (Gastrointestinal disorders) | 7 (7) | 0 (0) | 7 (7)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3)
Vomiting (Gastrointestinal disorders) | 2 (2) | 5 (5) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 3 (3) | 4 (4)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (3)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4)
Urinary tract infection (Gastrointestinal disorders) | 8 (9) | 13 (14) | 9 (10)
Coronavirus infection (Infections and infestations) | 11 (11) | 10 (11) | 6 (8)
Upper respiratory tract infection (Infections and infestations) | 5 (5) | 2 (2) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2) | 4 (4) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 4 (4) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1) | 3 (3) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 4 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 5 (5)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4) | 3 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 3 (3)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 7 (7) | 3 (3)
Diabetes mellitus (Metabolism and nutrition disorders) | 6 (6) | 3 (3) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 3 (3)
Procedural pain (Injury, poisoning and procedural complications) | 6 (7) | 4 (4) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 3 (3) | 2 (2)
Skin laceration (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 3 (3) | 0 (0) | 0 (0)
Low-density lipoprotein increased (Investigations) | 4 (4) | 3 (3) | 2 (2)
Coronavirus test positive (Investigations) | 1 (1) | 4 (4) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 4 (5) | 2 (3) | 0 (0)
Glycosylated hemoglobin increased (Investigations) | 1 (1) | 4 (4) | 0 (0)
Weight increased (Investigations) | 2 (2) | 0 (0) | 3 (3)
Headache (Nervous system disorders) | 7 (10) | 4 (5) | 6 (7)
Rash (Skin and subcutaneous tissue disorders) | 1 (3) | 3 (5) | 3 (4)
Fatigue (General disorders) | 4 (4) | 4 (4) | 3 (3)
Edema peripheral (General disorders) | 3 (3) | 3 (3) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (6) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 3 (3) | 3 (3)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 3 (3)
Hypertension (Vascular disorders) | 4 (5) | 0 (0) | 4 (5)
Lymphadenopathy (Blood and lymphatic system disorders) | 4 (4) | 2 (2) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 2 (3) | 1 (1) | 3 (3)
Seasonal allergy (Immune system disorders) | 2 (2) | 3 (3) | 2 (2)
Hypothyroidism (Endocrine disorders) | 0 (0) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Each Investigator is obligated to keep data pertaining to the study confidential. The Investigator must consult with the Sponsor before any study data are submitted for publication. The Sponsor reserves the right to deny publication rights until mutual agreement on the content, format, interpretation of data in the manuscript, and journal selected for publication are achieved.

DOCUMENTS (2):
  • Study Protocol (2022-07-21): https://cdn.clinicaltrials.gov/large-docs/16/NCT04052516/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT04052516/SAP_001.pdf